CLINICAL TRIAL: NCT00720486
Title: Anger Management Treatment for Female Juvenile Offenders
Brief Title: Effectiveness of Anger Management Treatment in Reducing Anger-Related Behaviors in Female Juvenile Offenders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: naomi goldstein (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, naomi goldstein, PI, Drexel University
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH070400 (NIH); K23MH070400 (NIH); DSIR 82-SEMS
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Anger
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive Juvenile Justice Anger Management for Girls plus treatment as usual.
  Interventions: Behavioral: Juvenile Justice Anger Management (JJAM) for Girls; Behavioral: Treatment as usual
- 2 (Active Comparator): Participants will receive treatment as usual.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Juvenile Justice Anger Management (JJAM) for Girls — JJAM will include two 1.5-hour group treatment sessions per week for 8 weeks. JJAM sessions will be manual based and will be designed to help youth develop skills in the following areas: identifying different types of physical and relational aggression, recognizing early warning signs of anger, avoiding anger-provoking situations, managing anger to prevent aggression, solving problems, communicating about anger-related events, and repairing relationships damaged by anger-related behaviors.
  Arms: 1
Behavioral: Treatment as usual — Treatment as usual will include standard activities in the female juvenile justice program.

SUMMARY:
This study will evaluate the effectiveness of an anger management treatment program, Juvenile Justice Anger Management for Girls, in reducing anger-related behaviors displayed by girls in the juvenile justice system.

DETAILED DESCRIPTION:
Girls represent a growing segment of the juvenile justice population in the United States, with a large number of them being victims of sexual, physical, and psychological abuse. These girls have special needs in terms of treatment and rehabilitation; however, little research exists on effective mental health treatments for female juvenile offenders in justice facilities. Despite the severity of anger-related behaviors displayed by girls in the juvenile justice system, no anger management treatments have been systematically developed to meet the unique treatment needs of delinquent girls. Treatment programs that provide gender-specific education, counseling, and emotional support are necessary for addressing the aggressive behaviors and psychological distress often displayed among this population. One such treatment program, the Juvenile Justice Anger Management (JJAM) for Girls, is an anger management program adapted from Lochman's Coping Power program, an empirically supported school-based anger management treatment for younger children. This study will evaluate the effectiveness of JJAM for Girls in reducing anger-related behaviors displayed by girls in the juvenile justice system.

Participation in this study will last about 8 months. All participants will first undergo initial assessments that will include a combination of structured interviews, self-report measures, rating scales, and reviews of program behavioral records and incident reports. Participants will then be assigned randomly to receive JJAM for Girls plus treatment as usual or treatment as usual alone. Participants receiving JJAM for Girls will attend two 1.5-hour sessions per week for 8 weeks. Sessions will aim to help youth develop skills in the following areas: identifying different types of physical and relational aggression, recognizing early warning signs of anger, avoiding anger-provoking situations, managing anger to prevent aggression, solving problems, communicating about anger-related events, and repairing relationships damaged by anger-related behaviors. Participants will also complete between-session practice activities that will include practicing skills involved in planning personal goals. Treatment as usual for all participants will include all standard activities in the female juvenile justice program. All participants will repeat the initial assessments at treatment completion and Month 6 of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to one of the designated juvenile justice facilities
* Has the ability to speak, read, and understand English sufficiently well to complete the procedures of the study
* Disposition to the juvenile justice program must last the 8 weeks of scheduled treatment plus 1 week before and after treatment

Exclusion Criteria:

* Fails to complete pretreatment assessments
* Current psychotic symptoms, mental retardation, or severe developmental disabilities
* Considered to be a ward of the state (defined as a youth without a parent, either biological or adoptive, as the legal custodian)

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in anger | Measured at pretreatment, post-treatment, and Month 6 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Goldstein, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Goldstein NE, Kemp KA, Leff SS, Lochman JE. Guidelines for Adapting Manualized Interventions for New Target Populations: A Step-Wise Approach Using Anger Management as a Model. Clin Psychol (New York). 2012 Dec 1;19(4):385-401. doi: 10.1111/cpsp.12011. PMID 25110403
- [Background] Goldstein NE, Serico JM, Riggs Romaine CL, Zelechoski AD, Kalbeitzer R, Kemp K, Lane C. Development of the Juvenile Justice Anger Management Treatment for Girls. Cogn Behav Pract. 2013 May;20(2):171-188. doi: 10.1016/j.cbpra.2012.06.003. PMID 27642247
- [Background] Lane C, Goldstein NE, Heilbrun K, Cruise KR, Pennacchia D. Obstacles to research in residential juvenile justice facilities: recommendations for researchers. Behav Sci Law. 2012 Jan-Feb;30(1):49-68. doi: 10.1002/bsl.1991. Epub 2012 Jan 4. PMID 22298128